CLINICAL TRIAL: NCT02053519
Title: Can Vitamin D Supplementation Improve Hepatitis C Cure Rates : A Pilot Multicentre Randomised Controlled Clinical Trial
Brief Title: Can Vitamin D Supplementation Improve Hepatitis C Cure Rates
Acronym: ViaDUCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, John Dillon, Professor of Hepatology and Gastroenterology, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012GA03; 2013-003573-10 (EudraCT Number)
Record Dates: First submitted 2014-01-16; First posted 2014-02-03 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vigantol Oil, (Vitamin D3) (Active Comparator): Oral Vigantol Oil 5 mls, (100 000 iu of Vitamin D). First dose at randomisation, 7 -28 days prior to commencing standard Hepatitis C treatment for Hepatitis C Genotypes 1 or 3 . Thereafter monthly with concurrent Hepatitis C treatment.
  Interventions: Drug: Active Comparator: Vigantol Oil (Vitamin D3)
- MyGliol Oil (Placebo Comparator): Matched placebo. Subjects randomised to this arm will take 5 mls of active Placebo, (Mygliol oil), 7 - 28 days prior to commencing active Hepatitis C treatment and thereafter 5 mls monthly concurrent with Hepatitis C treatment for the duration of the study
  Interventions: Drug: Mygliol Oil

INTERVENTIONS:
Drug: Active Comparator: Vigantol Oil (Vitamin D3) — Vitamin D Oral oil 100.000iu in 5 mls
  Arms: Vigantol Oil, (Vitamin D3)
Drug: Mygliol Oil — Matched placebo comparator
  Arms: MyGliol Oil

SUMMARY:
Evidence suggests that vitamin D may be directly or indirectly a co-factor for the efficacy of Hepatitis C virus, (HCV), antiviral therapies. The level of vitamin D necessary for optimum immune function is ill defined and many of those with HCV infection in Scotland are below these levels. Vitamin D is a cheap and safe medication, so its addition to anti-viral therapy should be highly cost-effective even if only a modest increase in SVR was achieved. Given the Scottish HCV epidemic, the world leading government response to it and the nationally low vitamin D levels, Scotland is perfectly placed to answer this question. Therefore the investigators hypothesize that vitamin D supplementation will improve SVR and propose a randomised controlled trial to test this hypothesis. The anticipated end of study date for this study is April 2015

DETAILED DESCRIPTION:
Hepatitis C is a major health problem for Scotland with greater than 1% of the population infected; the Scottish Government has recognised this and mounted the Hepatitis C action plan, recognised as the world leading public health response to the epidemic. The key aim of this is to expand treatment access and numbers of patients cured of HCV infection to prevent patients developing the complications of cirrhosis and hepatocellular carcinoma.

The success of treatment for HCV depends on genotype and is measured by the Sustained Viral Response (SVR). The SVR is the absence of virus 24 weeks after end of treatment and has been shown to be a cure of infection. The FDA has recently suggested SVR can be assessed at 12 weeks, in clinical trials. Scotland has an equal mix of genotype 1 & 3 HCV infection accounting for greater than 95% of those infected. Treatment involves Pegylated Interferon injections weekly and Ribavirin twice daily for 6 months for HCV genotype 3 infection, with an SVR of 70%. For genotype 1 infection treatment is with the above dual therapy with the addition of a protease inhibitor, for treatment duration of 6-12 months leading to SVR rates of 65-70%. There are an increasing number of new pharmacological products in advanced development that will be available for clinicians to use but these, as well as increasing efficacy, will increase cost. So it requires clinicians to make treatment as effective as possible.

Vitamin D has traditionally been associated with bone health, with definite deficiency causing osteomalacia and making a contribution to osteoporosis. The traditional, currently used normal ranges for Vitamin D are based on prevention of bone diseases. Recently and controversially it has been suggested that low normal levels of vitamin D are associated with multiple other disease states, including cancer, infection and cardiovascular disease Additionally it has been suggested that many of the normal population in Scotland are vitamin D deficient. Other studies have shown that drug users, a high risk group for HCV infection have similarly deficient levels of vitamin D. Studies have suggested that up to 92% of those with chronic liver disease have vitamin D levels below that deemed acceptable physiologically to maintain health.

Some data is now available to support the role of vitamin D supplementation in the treatment of hepatitis C and improving SVR rates. Several observational studies have found an association between low vitamin D levels and reduced SVR rates, and additionally one study has shown an association between a single nucleotide polymorphism (SNP) in vitamin D binding protein and treatment response. A small Israeli trial of vitamin D supplementation in HCV treatment has shown increased SVRs in those supplemented, but the study had a number of flaws including a failure of randomisation(13). Additionally there have been an abstract and a letter report of improved outcome with a vitamin D intervention . Biological mechanisms of interaction between vitamin D and the immune system have been explored. It has been shown that Vitamin D plays a role in the regulation of innate immunity, macrophage function, and cell mediated immunity Vitamin D receptors (VDR) are also expressed on many effector cells of the immune system; activated T and B cells, macrophages and monocytes which act to increase to enhance phagocytic action and interferon activity , it has also been suggested vitamin D has a direct effect on HCV. These give a biological basis for the effect of vitamin D on the success of antiviral therapy.

A randomised controlled trial, to be successful, requires recruitment and retention of subjects in the trial. HCV infection is associated with chaotic lifestyles which might impair the rate of recruitment and retention, although the Scottish HCV clinical database audit clearly shows that, with all comers, routine HCV care in Scotland matches the results from the randomised clinical trials. This pilot study will also help determine the recruitment and retention rates for a larger trial in this population.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible if they

* Have confirmed hepatitis C with positive PCR for genotype 1 or 3
* Are planned to commence on standard eradication therapy for HCV
* Aged 18 or over

Exclusion Criteria:

* Exclusion criteria are:

  * Hepatitis C genotype other than 1 or 3
  * Contraindications to interferon / ribavirin therapy
  * eGFR <30 ml/min (by MDRD4 method)
  * Currently decompensated liver disease

    o Ascites, encephalopathy or variceal bleeding
  * History of renal calculi
  * Serum calcium <2.15 mmol/L or >2.60 mmol/L
  * History of sarcoidosis, metastatic malignancy
  * Hepatocellular carcinoma (current or previous)
  * Taking >400 units/day of vitamin D
  * HIV positive
  * Pregnancy
  * Breastfeeding
  * Of childbearing potential and not taking reliable contraception
  * Unable to provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the number of patients with sustained virologic responses, (SVR), at 12 weeks post standard therapy on Vitamin D3 as compared to placebo | at 12 weeks and at12 months
  viral response by Polymerase Chain Reaction, (PCR), will be measured at 12 weeks of treatment and then again at 12 months, (24 weeks following treatment) to measure response to treatment and assess in how many participants this is sustained at 24 weeks following treatment, (ie 12 months)

SECONDARY OUTCOMES:
Secondary Objectives | Assessed at week 4, week 12 and week 24 of the Clinical Trial
  • The number of patients with rapid virological response (RVR is defined as negative Hepatitis C Virus Polymerase Chain Reaction, (HCV PCR), at 4 weeks of therapy) and who therefore receive response guided shortened therapy.

CONTACTS AND LOCATIONS:
Overall Officials: John Dillon, MD, Principal Investigator — University of Dundee
Locations (6):
- United Kingdom (6):
  - NHS Grampian, Aberdeen
  - NHS Tayside, Dundee
  - NHS Lothian, Edinburgh
  - NHS Forth Valley, Falkirk
  - NHS Greater Glasgow and Clyde, Glasgow
  - NHS Greater Glasgow and Clyde, Paisley